CLINICAL TRIAL: NCT00498680
Title: A Prospective, Randomized, 3-arm Parallel Trial to Evaluate the Safety and Clinical Effectiveness of 2 Lower Dose Combined PDE5i's vs. Single Maximal Dose PDE5i Treatment
Brief Title: Safety and Clinical Effectiveness of 2 Lower Dose Combined PDE5i's vs. Single Maximal Dose PDE5i
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Prof. Vardi Yoram, RAMBAM HEALTH CARE CAMPUS
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2431-ctil
Record Dates: First submitted 2007-07-08; First posted 2007-07-10 (Estimated); Last update posted 2010-10-22 (Estimated); Status verified 2007-01

CONDITIONS: Impotence
Keywords: Erectile Dysfunction; Treatment; PDE5i
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate; Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Viagra 100mg (Active Comparator)
  Interventions: Drug: Sildenafil
- Levitra 20mg (Active Comparator)
  Interventions: Drug: Vardenafil
- Viagra 50mg+ Levitra 10mg (Active Comparator)
  Interventions: Drug: Sildenafil, Vardenafil; Drug: Sildenafil & Vardenafil

INTERVENTIONS:
Drug: Sildenafil, Vardenafil — Sildenafil 100mg, vardenafil 20mg, combination of both half dosage.
  Other Names: Viagra, Levitra
  Arms: Viagra 50mg+ Levitra 10mg
Drug: Sildenafil — 100mg
  Arms: Viagra 100mg
Drug: Vardenafil — 20mg
  Arms: Levitra 20mg
Drug: Sildenafil & Vardenafil — 50mg & 10 mg
  Arms: Viagra 50mg+ Levitra 10mg

SUMMARY:
A prospective, randomized, 3-arm parallel trial on 45 males with ED that were never exposed to PDE5i therapy (naïve patients) will be enrolled.In each group, every patient will receive three treatment regimes (Viagra®50mg & Levitra®10mg, Viagra®100mg, Levitra®20mg), in different sequences of administration in such a manner that eventually each patient will receive all regimes in a double- blinded fasion.Safety will be evaluated at pre- screening by measuring hourly vital signs (blood pressure, heart rate)for 4 consecutive hours after taking half-dose combination. Any decrease in blood pressure of 20 mmhg below baseline will exclude the subject from the study. Effcacy will be evaluated by questionnaires (IIEF, Quality of erection questionnaire, grade of erection scale, Sear, QVS and Sexual Encounter Profiles for each sexual event). Non-parametric statistical analysis of the collected data Comparing the 3 groups will be performed.

DETAILED DESCRIPTION:
A prospective, randomized, 3-arm parallel trial on 45 males with ED that were never exposed to PDE5i therapy (naïve patients) will be enrolled. Recruitment will be performed via advertisement or by offering newly diagnosed naïve ED patients visiting the clinic to participate in the study.

In each group, every patient will receive three treatment regimes (Viagra®50mg & Levitra®10mg, Viagra®100mg, Levitra®20mg), in different sequences of administration, as follows:

Group 1) 15 naïve patients will start with Viagra®100mg, continue with Levitra®20mg and end the study with combined Viagra®50mg & Levitra®10mg.

Group 2) 15 naïve patients will start with combined Viagra®50mg & Levitra®10mg, continue with Levitra®20mg and end the study with Viagra®100mg.

Group 3) 15 naïve patients will start with Levitra®20mg, continue with Viagra®100mg and end the study with combined Viagra®50mg & Levitra®10mg.

Inclusion criteria: - Relationship with the same partner for at least 3 month

* Age ranging between 35-65 years old
* Sexually active, (minimal frequency of one sexual encounter per 2 weeks)
* IIEF ED domain score 22 and below. Exclusion criteria: - Subjects with premature ejaculation as their main sexual complaint.
* Subjects with severe cardiovascular disease in the past 6 months, including cardiac failure, myocardial infarction, unstable angina, stroke or transient ischemic attack, symptomatic or clinically significant cardiac arrhythmias including atrial fibrillation,
* Subjects with Contraindications to PDE5i therapy. Namely patients receiving treatment with nitrate based medication or patients that for various reasons cannot take PDE5 inhibitors (severe hepatic diseases- cirrhosis or ALT (Alanine aminotransferase)>2x upper limit of normal), renal impairment (creatinine clearance > 30ml/min) or known hereditary degenerative retinal disorders such as retinitis pigmentosa. ,
* Concomitant treatment with potent CYP3A4 and CYP2C9 inhibitors (e.g protease inhibitors ritonavir and saquinavir, ketoconazole, itrakonazole, miconazole, nefazodone, claritromycin, troleandomycin, erythromycin and cimetidine)
* Subjects mentally unfit for the study.

SAFETY & ELIGIBILITY VISIT. After a thorough explanation of the nature of the study and its protocol and after understanding and signing the informed consent form. In this visit, each subject will start the study by measuring basic blood pressure levels and pulse rate. Under our supervision the subject will take the combined half dose as suggested. Blood pressure monitoring and pulse rate every half- hour at the clinic will be performed for 4 hours (according to the pharmacokinetic properties of the medications) . Any recordings of 20 mmhg below baseline will exclude the subject from the study. If no significant effect on blood pressure will be noted, the subject will be eligible for inclusion in the study, and will be invited for the FIRST visit 7 days later. ( a washout period of one week is sufficient to eliminate any effect of one-time dosing of the combined half dose treatment). Each included patient in the coming 6 visits will respond to the following pre-set sexual function and satisfaction questionnaires (Hebrew validated):

1. The full IIEF (International Index Erectile Function) standard Questionnaire
2. The SEAR (Self-Esteem And Relationship) questionnaire
3. QVS (Quality of Sexual Life) questionnaire
4. Quality of erection questionnaire
5. Grade of erection scale

At each visit, documentation of side-effects will be done and a physical examination (blood pressure and pulse rate) will be done. A 24 hour mobile phone dedicated to patient inquiries will be provided to each patient during the whole study.

Visit 1: The subject will be offered, at random, for 4 attempts at home, either a combination dose regime (Viagra®50mg & Levitra®10mg, 4 tablets each) or 4 tablets of Viagra®100mg single dose or 4 tablets of Levitra® 20 mg. The subject will also receive 6 SEP (Sexual Encounter Profile) diaries to fill out at home after each sexual attempt. After 4 attempts the subject will return for visit 2, will respond to the same questionnaires and an additional EDITS (Erectile Dysfunction Inventory of Treatment Satisfaction) questionnaire. A new visit will be rescheduled for 2 weeks later to allow a washout period. At visit 3 they will receive the 2nd regime and 4 new SEP diaries, and after 4 attempts will return to visit 4, fill out the same 4 questionnaires. Again, a new visit will be rescheduled for 2 weeks later to allow a washout period. On visit 5 they will return to receive the third treatment regime. Again, they will receive 4 SEP diaries to fill out after each sexual attempt at home. At their final visit (visit 6), in addition to the other 4 questionnaires, the patients will be required to respond to a preference questionnaire regarding the preferred regime.

The approximate timeline for performing the study for every patient is 1/2 a year from recruitment. The estimated timeline for completion of the study is 16 months.

*Only on inclusion

** Washout period 2 weeks

Non-parametric statistical analysis of the collected data from the questionnaires will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Relationship with the same partner for at least 3 month
* Age ranging between 35-65 years old
* Sexually active, (minimal frequency of one sexual encounter per 2 weeks)
* IIEF ED domain score 22 and below.

Exclusion Criteria:

* Subjects with premature ejaculation as their main sexual complaint.
* Subjects with severe cardiovascular disease in the past 6 months, including cardiac failure, myocardial infarction, unstable angina, stroke or transient ischemic attack, symptomatic or clinically significant cardiac arrhythmias including atrial fibrillation,
* Subjects with Contraindications to PDE5i therapy. Namely patients receiving treatment with nitrate based medication or patients that for various reasons cannot take PDE5 inhibitors (severe hepatic diseases- cirrhosis or ALT (Alanine aminotransferase)>2x upper limit of normal), renal impairment (creatinine clearance > 30ml/min) or known hereditary degenerative retinal disorders such as retinitis pigmentosa. ,
* Concomitant treatment with potent CYP3A4 and CYP2C9 inhibitors (e.g protease inhibitors ritonavir and saquinavir, ketoconazole, itrakonazole, miconazole, nefazodone, claritromycin, troleandomycin, erythromycin and cimetidine)
* Subjects mentally unfit for the study.

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2007-03; Primary Completion 2011-01 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
increase of 5 points or more in the IIEF erectile function domain | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Ilan Gruenwald, MD, Principal Investigator — Israel Urology Association
Locations (1):
- Neuro-urology unit, Rambam Medical Center, Haifa, Israel